CLINICAL TRIAL: NCT00471081
Title: Study to Assess Immunogenicity, Reactogenicity and Safety of Primary Vaccination With GSK Biologicals' MenACWY Vaccine (GSK134612) Given as 1 or 2 Doses to Healthy Toddlers 9-12 Months of Age
Brief Title: Immunogenicity and Safety of Meningococcal Vaccine GSK134612 Given as 1 or 2 Doses to Healthy 9-12 Months Old Toddlers.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109375
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Infections, Meningococcal
Keywords: Neisseria meningitidis;; Humans;; Meningococcal vaccines;; Safety; Vaccines, conjugate;; Toddlers;; Immunogenicity;
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Group A (Experimental): Single dose GSK134612.
  Interventions: Biological: Meningococcal vaccine GSK134612
- Group B (Experimental): Two doses of GSK134612.
  Interventions: Biological: Meningococcal vaccine GSK134612

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — One or 2 intramuscular injections.

SUMMARY:
The purpose of the study is to characterize the safety and immunogenicity of 1 dose of GSK134612 vaccine at 12 months of age and of GSK134612 vaccine administered as 2 doses at 9 and 12 months of age.

DETAILED DESCRIPTION:
The protocol posting has been amended to reflect changes as a consequence of an amendment to the protocol and also to comply with the FDA amendment Act, Sep 2007. Sections impacted are Brief Title, Official Title of the study, Brief Summary, Key Inclusion & Exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose parents/guardians the investigator believes can and will comply with the requirements of the protocol
* A male or female of 9 months of age (has not attained 10 months of age) at the time of enrollment.
* Up to date on vaccinations based on ACIP recommendations and the standard practice at the investigational site.
* Written informed consent obtained from parents/guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding enrollment, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 1 month of a dose of study vaccine(s), with the exception of influenza vaccine.
* Planned administration of a tetanus toxoid (TT) containing vaccine throughout the active phase of the study (through one month after the last vaccination).
* Previous vaccination with meningococcal polysaccharide or conjugate vaccine of serogroup A, C W and/or Y.
* History of meningococcal diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination (no laboratory testing is required).
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrollment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the active phase of the study (through one month after the last dose of study vaccine).

Ages: 9 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 385 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2008-10-23 (Actual); Study Completion 2008-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- United States (18):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Antioch, California
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Madera, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Vacaville, California
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Westminster, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Birmingham, Georgia
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Amarillo, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Klein NP, Baine Y, Bianco V, Lestrate PR, Naz A, Blatter M, Friedland LR, Miller JM. One or two doses of quadrivalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine is immunogenic in 9- to 12-month-old children. Pediatr Infect Dis J. 2013 Jul;32(7):760-7. doi: 10.1097/INF.0b013e31828693c5. PMID 23348814
- [Background] Klein N et al. Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal ACWY Tetanus Toxoid Conjugate Vaccine in Healthy Toddlers: 1-year Persistence. Abstract presented at the 51st Annual Interscience Conference on Antimicrobial Agents & Chemotherapy. Chicago, US, 17-20 September 2011.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 109375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109375 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 196 subjects were enrolled and randomized in the GSK 134612 1 dose Group at the study start but 36 subjects were not vaccinated, due to the 3-month period between enrollment and vaccination.
Pre-assignment Details: The majority of subjects withdrawn in the active Phase were still contacted for the safety follow-up, therefore the subjects listed as withdrawn were not necessarily the same individuals in the two phases (Active Phase and Extended Safety Follow-Up).
Groups:
- GSK 134612 1 Dose Group: Healthy male or female subjects of 9 months of age at the time of enrollment received 1 dose of GSK 134612 vaccine at 12 months of age, administered intramuscularly in the left thigh.
- GSK 134612 2 Doses Group: Healthy male or female subjects of 9 months of age at the time of enrollment received 1 dose of GSK 134612 at 9 months of age and another dose at 12 months of age, administered intramuscularly in the left thigh.
Period: Active Phase
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Started | 160 | 189
Completed | 158 | 176
Not Completed | 2 | 13
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lost health plan/insurance | 1 | 8
Period: Extended Safety Follow-Up
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Started | 160 | 189
Completed | 158 | 176
Not Completed | 2 | 13
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 8
Not completed — Missing confirmed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group | Total
Number analyzed (Participants) | 160 | 189 | 349
Age, Continuous [Mean (Standard Deviation); unit: Months] | 9 (0.08) | 9 (0.0) | 9 (0.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 101 | 178
  Male | 83 | 88 | 171

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serum Bactericidal Assay Using Human Complement Against Neisseria Meningitides Serogroups A, C, W-135, Y (hSBA-MenA, hSBA-MenC, hSBA-MenW -135 and hSBA-Men-Y) Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:8.
Time Frame: One month after the last dose (at Month 4)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 132 | 146
Participants
  hSBA-MenA: number analyzed (Participants) | 132 | 138
  hSBA-MenA | 105 | 122
  hSBA-MenC: number analyzed (Participants) | 130 | 137
  hSBA-MenC | 123 | 137
  hSBA-MenW-135: number analyzed (Participants) | 118 | 143
  hSBA-MenW-135 | 60 | 142
  hSBA-MenY | 74 | 145
Statistical Analysis 1: Comparison: GSK 134612 2 Doses Group; To demonstrate the immunogenicity of GSK134612 administered on a 2-dose schedule at 9 and 12 months of age with respect to serum bactericidal assay using human complement (hSBA) titers ≥1:8 for each discrete N. meningitidis serogroup A; Test type: Superiority; Percentage of subjects with hSBA titers = 88.4, 95% CI 2-sided [81.9 to 93.2] — Immunogenecity of GSK134612 was demonstrated if the lower limit (LL) of the 2-sided exact 95% confidence interval (CI) was higher than the pre-defined clinical limit of 80%
Statistical Analysis 2: Comparison: GSK 134612 2 Doses Group; To demonstrate the immunogenicity of GSK134612 administered on a 2-dose schedule at 9 and 12 months of age with respect to serum bactericidal assay using human complement (hSBA) titers ≥1:8 for each discrete N. meningitidis serogroup C; Test type: Superiority; Percentage of subjects with hSBA titers = 100, 95% CI 2-sided [97.3 to 100] — Immunogenecity of GSK134612 was demonstrated if the lower limit (LL) of the 2-sided exact 95% confidence interval (CI) was higher than the pre-defined clinical limit of 90%
Statistical Analysis 3: Comparison: GSK 134612 2 Doses Group; To demonstrate the immunogenicity of GSK134612 administered on a 2-dose schedule at 9 and 12 months of age with respect to serum bactericidal assay using human complement (hSBA) titers ≥1:8 for each discrete N. meningitidis serogroup W-135; Test type: Superiority; Percentage of subjects with hSBA titers = 99.3, 95% CI 2-sided [96.2 to 100] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: GSK 134612 2 Doses Group; To demonstrate the immunogenicity of GSK134612 administered on a 2-dose schedule at 9 and 12 months of age with respect to serum bactericidal assay using human complement (hSBA) titers ≥1:8 for each discrete N. meningitidis serogroup Y; Test type: Superiority; Percentage of subjects with hSBA titers = 99.3, 95% CI 2-sided [96.2 to 100] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay Using hSBA-MenA, hSBA-MenC, hSBA-MenW -135 and hSBA-Men-Y Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:8.
Time Frame: One month after the first dose (at Month 1)
Population: This analysis was performed on subjects who have received the Month 0 vaccination in the GSK 134612 2 doses Group from the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 131
Participants
  hSBA-MenA: number analyzed (Participants) | 128
  hSBA-MenA | 81
  hSBA-MenC: number analyzed (Participants) | 127
  hSBA-MenC | 115
  hSBA-MenW-135: number analyzed (Participants) | 117
  hSBA-MenW-135 | 22
  hSBA-MenY | 49

3. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay Using hSBA-MenA, hSBA-MenC, hSBA-MenW -135 and hSBA-Men-Y Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the hSBA titers was greater than or equal to (≥) 1:4.
Time Frame: At Month 1 (for GSK 134612 2 doses Group only) and Month 4
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available. Month 1 data are not available for the GSK 134612 1 dose Group (only vaccinated at Month 3).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 132 | 146
Participants
  hSBA-MenA, Month 1: number analyzed (Participants) | 0 | 128
  hSBA-MenA, Month 1 |  | 90
  hSBA-MenA, Month 4: number analyzed (Participants) | 132 | 138
  hSBA-MenA, Month 4 | 115 | 122
  hSBA-MenC, Month 1: number analyzed (Participants) | 0 | 127
  hSBA-MenC, Month 1 |  | 115
  hSBA-MenC, Month 4: number analyzed (Participants) | 130 | 137
  hSBA-MenC, Month 4 | 123 | 137
  hSBA-MenW-135, Month 1: number analyzed (Participants) | 0 | 117
  hSBA-MenW-135, Month 1 |  | 24
  hSBA-MenW-135, Month 4: number analyzed (Participants) | 118 | 143
  hSBA-MenW-135, Month 4 | 63 | 142
  hSBA-MenY, Month 1: number analyzed (Participants) | 0 | 131
  hSBA-MenY, Month 1 |  | 52
  hSBA-MenY, Month 4 | 79 | 145

4. Secondary Outcome: hSBA-MenA, hSBA-MenC, hSBA-MenW -135 and hSBA-Men-Y Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Month 1 (for GSK 134612 2 doses Group only) and Month 4
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 132 | 146
Titers
  hSBA-MenA, Month 1: number analyzed (Participants) | 0 | 128
  hSBA-MenA, Month 1 |  | 13.6 [10.5 to 17.7]
  hSBA-MenA, Month 4: number analyzed (Participants) | 132 | 138
  hSBA-MenA, Month 4 | 24.9 [19.5 to 31.9] | 50.8 [39.6 to 65.1]
  hSBA-MenC, Month 1: number analyzed (Participants) | 0 | 127
  hSBA-MenC, Month 1 |  | 83.7 [63.8 to 110.0]
  hSBA-MenC, Month 4: number analyzed (Participants) | 130 | 137
  hSBA-MenC, Month 4 | 161.5 [126.3 to 206.5] | 1105.5 [906.2 to 1348.6]
  hSBA-MenW-135, Month 1: number analyzed (Participants) | 0 | 117
  hSBA-MenW-135, Month 1 |  | 3.5 [2.8 to 4.3]
  hSBA-MenW-135, Month 4: number analyzed (Participants) | 118 | 143
  hSBA-MenW-135, Month 4 | 11.6 [8.2 to 16.4] | 1062.9 [878.4 to 1286.3]
  hSBA-MenY, Month 1: number analyzed (Participants) | 0 | 131
  hSBA-MenY, Month 1 |  | 7.0 [5.2 to 9.5]
  hSBA-MenY, Month 4 | 15.7 [11.1 to 22.1] | 475.2 [392.2 to 575.9]

5. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay Using Rabbit Complement Against Neisseria Meningitides Serogroups A, C, W-135, Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY) Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8.
Time Frame: At Month 1 (for GSK 134612 2 doses Group only) and Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 51 | 51
Participants
  rSBA-MenA, Month 1: number analyzed (Participants) | 0 | 41
  rSBA-MenA, Month 1 |  | 41
  rSBA-MenA, Month 4: number analyzed (Participants) | 51 | 47
  rSBA-MenA, Month 4 | 51 | 47
  rSBA-MenC, Month 1: number analyzed (Participants) | 0 | 43
  rSBA-MenC, Month 1 |  | 42
  rSBA-MenC, Month 4 | 51 | 51
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 0 | 43
  rSBA-MenW-135, Month 1 |  | 43
  rSBA-MenW-135, Month 4: number analyzed (Participants) | 51 | 50
  rSBA-MenW-135, Month 4 | 51 | 50
  rSBA-MenY, Month 1: number analyzed (Participants) | 0 | 42
  rSBA-MenY, Month 1 |  | 42
  rSBA-MenY, Month 4: number analyzed (Participants) | 50 | 50
  rSBA-MenY, Month 4 | 50 | 50

6. Secondary Outcome: Number of Subjects With Serum Bactericidal Assay Using rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Antibody Titers Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:128.
Time Frame: At Month 1 (GSK 134612 2 doses Group only) and Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 51 | 51
Participants
  rSBA-MenA, Month 1: number analyzed (Participants) | 0 | 41
  rSBA-MenA, Month 1 |  | 41
  rSBA-MenA, Month 4: number analyzed (Participants) | 51 | 47
  rSBA-MenA, Month 4 | 50 | 47
  rSBA-MenC, Month 1: number analyzed (Participants) | 0 | 43
  rSBA-MenC, Month 1 |  | 35
  rSBA-MenC, Month 4 | 44 | 50
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 0 | 43
  rSBA-MenW-135, Month 1 |  | 43
  rSBA-MenW-135, Month 4: number analyzed (Participants) | 51 | 50
  rSBA-MenW-135, Month 4 | 51 | 50
  rSBA-MenY, Month 1: number analyzed (Participants) | 0 | 42
  rSBA-MenY, Month 1 |  | 42
  rSBA-MenY, Month 4: number analyzed (Participants) | 50 | 50
  rSBA-MenY, Month 4 | 49 | 50

7. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW -135 and rSBA-Men-Y Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Month 1 (GSK 134612 2 doses Group only) and Month 4
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 51 | 51
Titers
  rSBA-MenA, Month 1: number analyzed (Participants) | 0 | 41
  rSBA-MenA, Month 1 |  | 1092.6 [839.0 to 1422.9]
  rSBA-MenA, Month 4: number analyzed (Participants) | 51 | 47
  rSBA-MenA, Month 4 | 1911.5 [1390.1 to 2628.5] | 1179.1 [931.0 to 1493.3]
  rSBA-MenC, Month 1: number analyzed (Participants) | 0 | 43
  rSBA-MenC, Month 1 |  | 229.3 [165.4 to 317.9]
  rSBA-MenC, Month 4 | 456.3 [336.2 to 619.4] | 1484.4 [1110.3 to 1984.6]
  rSBA-MenW-135, Month 1: number analyzed (Participants) | 0 | 43
  rSBA-MenW-135, Month 1 |  | 1412.3 [1029.7 to 1936.9]
  rSBA-MenW-135, Month 4: number analyzed (Participants) | 51 | 50
  rSBA-MenW-135, Month 4 | 3069.9 [2246.9 to 4194.4] | 1771.6 [1363.0 to 2302.7]
  rSBA-MenY, Month 1: number analyzed (Participants) | 0 | 42
  rSBA-MenY, Month 1 |  | 817.1 [671.0 to 995.1]
  rSBA-MenY, Month 4: number analyzed (Participants) | 50 | 50
  rSBA-MenY, Month 4 | 1521.0 [1100.8 to 2101.7] | 1125.9 [938.7 to 1350.3]

8. Secondary Outcome: Number of Subjects With Anti-polysaccharide Meningococcal Serogroup A (Anti-PSA), Serogroup C (Anti-PSC), Serogroup W-135 (Anti-PSW-135) and Serogroup Y (Anti-PSY) Antibody Concentrations Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations was greater than or equal to (≥) 0.3 micrograms per milliliter (μg/mL).
Time Frame: At Month 1 (GSK 134612 2 doses Group only) and Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 60 | 66
Participants
  Anti-PSA, Month 1: number analyzed (Participants) | 0 | 35
  Anti-PSA, Month 1 |  | 35
  Anti-PSA, Month 4: number analyzed (Participants) | 26 | 29
  Anti-PSA, Month 4 | 26 | 29
  Anti-PSC, Month 1: number analyzed (Participants) | 0 | 66
  Anti-PSC, Month 1 |  | 66
  Anti-PSC, Month 4: number analyzed (Participants) | 60 | 56
  Anti-PSC, Month 4 | 60 | 56
  Anti-PSW-135, Month 1: number analyzed (Participants) | 0 | 31
  Anti-PSW-135, Month 1 |  | 31
  Anti-PSW-135, Month 4: number analyzed (Participants) | 31 | 54
  Anti-PSW-135, Month 4 | 30 | 54
  Anti-PSY, Month 1: number analyzed (Participants) | 0 | 25
  Anti-PSY, Month 1 |  | 25
  Anti-PSY, Month 4: number analyzed (Participants) | 36 | 46
  Anti-PSY, Month 4 | 36 | 46

9. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY Antibody Concentrations Greater Than or Equal to the Cut-off Value
Description: The cut-off value for the anti-polysaccharide concentrations was greater than or equal to (≥) 2.0 micrograms per milliliter (μg/mL).
Time Frame: At Month 1 (GSK 134612 s doses Group only) and Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 60 | 66
Participants
  Anti-PSA, Month 1: number analyzed (Participants) | 0 | 35
  Anti-PSA, Month 1 |  | 35
  Anti-PSA, Month 4: number analyzed (Participants) | 26 | 29
  Anti-PSA, Month 4 | 26 | 27
  Anti-PSC, Month 1: number analyzed (Participants) | 0 | 66
  Anti-PSC, Month 1 |  | 65
  Anti-PSC, Month 4: number analyzed (Participants) | 60 | 56
  Anti-PSC, Month 4 | 59 | 40
  Anti-PSW-135, Month 1: number analyzed (Participants) | 0 | 31
  Anti-PSW-135, Month 1 |  | 26
  Anti-PSW-135, Month 4: number analyzed (Participants) | 31 | 54
  Anti-PSW-135, Month 4 | 29 | 53
  Anti-PSY, Month 1: number analyzed (Participants) | 0 | 25
  Anti-PSY, Month 1 |  | 16
  Anti-PSY, Month 4: number analyzed (Participants) | 36 | 46
  Anti-PSY, Month 4 | 33 | 46

10. Secondary Outcome: Anti-PSC, Anti-PSW-135 and Anti-PSY Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL).
Time Frame: At Month 1 (GSK 134612 2 doses Group only) and Month 4
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 60 | 66
μg/mL
  Anti-PSA, Month 1: number analyzed (Participants) | 0 | 35
  Anti-PSA, Month 1 |  | 12.39 [9.31 to 16.48]
  Anti-PSA, Month 4: number analyzed (Participants) | 26 | 29
  Anti-PSA, Month 4 | 35.92 [25.68 to 50.23] | 5.59 [4.20 to 7.44]
  Anti-PSC, Month 1: number analyzed (Participants) | 0 | 66
  Anti-PSC, Month 1 |  | 8.15 [7.05 to 9.42]
  Anti-PSC, Month 4: number analyzed (Participants) | 60 | 56
  Anti-PSC, Month 4 | 10.91 [9.26 to 12.86] | 3.42 [2.85 to 4.09]
  Anti-PSW-135, Month 1: number analyzed (Participants) | 0 | 31
  Anti-PSW-135, Month 1 |  | 4.42 [3.20 to 6.11]
  Anti-PSW-135, Month 4: number analyzed (Participants) | 31 | 54
  Anti-PSW-135, Month 4 | 7.37 [4.89 to 11.12] | 13.47 [10.99 to 16.51]
  Anti-PSY, Month 1: number analyzed (Participants) | 0 | 25
  Anti-PSY, Month 1 |  | 3.40 [2.17 to 5.33]
  Anti-PSY, Month 4: number analyzed (Participants) | 36 | 46
  Anti-PSY, Month 4 | 8.19 [5.71 to 11.73] | 12.43 [9.95 to 15.53]

11. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) and 8-day (Days 0-7) periods following each vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects who had the symptoms sheet filled in and for whom data were available. Post-Dose 2 data are not available for the GSK 134612 1 dose Group (received a single vaccination).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 156 | 182
Participants
  Any Pain, Dose 1, Days 0-3 | 34 | 54
  Grade 3 Pain, Dose 1, Days 0-3 | 0 | 0
  Any Redness, Dose 1, Days 0-3 | 28 | 49
  Grade 3 Redness, Dose 1, Days 0-3 | 0 | 1
  Any Swelling, Dose 1, Days 0-3 | 13 | 27
  Grade 3 Swelling, Dose 1, Days 0-3 | 1 | 1
  Any Pain, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Any Pain, Dose 2, Days 0-3 |  | 42
  Grade 3 Pain, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Grade 3 Pain, Dose 2, Days 0-3 |  | 1
  Any Redness, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Any Redness, Dose 2, Days 0-3 |  | 37
  Grade 3 Redness, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Grade 3 Redness, Dose 2, Days 0-3 |  | 0
  Any Swelling, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Any Swelling, Dose 2, Days 0-3 |  | 19
  Grade 3 Swelling, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Grade 3 Swelling, Dose 2, Days 0-3 |  | 0
  Any Pain, Dose 1, Days 0-7 | 35 | 54
  Grade 3 Pain, Dose 1, Days 0-7 | 0 | 0
  Any Redness, Dose 1, Days 0-7 | 28 | 49
  Grade 3 Redness, Dose 1, Days 0-7 | 0 | 1
  Any Swelling, Dose 1, Days 0-7 | 13 | 27
  Grade 3 Swelling, Dose 1, Days 0-7 | 1 | 1
  Any Pain, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Any Pain, Dose 2, Days 0-7 |  | 42
  Grade 3 Pain, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Grade 3 Pain, Dose 2, Days 0-7 |  | 1
  Any Redness, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Any Redness, Dose 2, Days 0-7 |  | 37
  Grade 3 Redness, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Grade 3 Redness, Dose 2, Days 0-7 |  | 0
  Any Swelling, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Any Swelling, Dose 2, Days 0-7 |  | 19
  Grade 3 Swelling, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Grade 3 Swelling, Dose 2, Days 0-7 |  | 0

12. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary, oral, tympanic or rectal temperature equal to or above (≥) 38 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever higher than (>) 40.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) and 8-day (Days 0-7) periods following each vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 157 | 184
Participants
  Any Drowsiness, Dose 1, Days 0-3 | 42 | 63
  Grade 3 Drowsiness, Dose 1, Days 0-3 | 1 | 0
  Related Drowsiness, Dose 1, Days 0-3 | 32 | 51
  Any Fever, Dose 1, Days 0-3 | 12 | 4
  Grade 3 Fever, Dose 1, Days 0-3 | 0 | 0
  Related Fever, Dose 1, Days 0-3 | 7 | 1
  Any Irritability, Dose 1, Days 0-3 | 63 | 101
  Grade 3 Irritability, Dose 1, Days 0-3 | 2 | 4
  Related Irritability, Dose 1, Days 0-3 | 48 | 87
  Any Loss of appetite, Dose 1, Days 0-3 | 34 | 42
  Grade 3 Loss of appetite, Dose 1, Days 0-3 | 1 | 1
  Related Loss of appetite, Dose 1, Days 0-3 | 19 | 31
  Any Drowsiness, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Any Drowsiness, Dose 2, Days 0-3 |  | 47
  Grade 3 Drowsiness, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Grade 3 Drowsiness, Dose 2, Days 0-3 |  | 0
  Related Drowsiness, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Related Drowsiness, Dose 2, Days 0-3 |  | 36
  Any Fever, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Any Fever, Dose 2, Days 0-3 |  | 11
  Grade 3 Fever, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Grade 3 Fever, Dose 2, Days 0-3 |  | 0
  Related Fever, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Related Fever, Dose 2, Days 0-3 |  | 4
  Any Irritability, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Any Irritability, Dose 2, Days 0-3 |  | 77
  Grade 3 Irritability, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Grade 3 Irritability, Dose 2, Days 0-3 |  | 3
  Related Irritability, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Related Irritability, Dose 2, Days 0-3 |  | 59
  Any Loss of appetite, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Any Loss of appetite, Dose 2, Days 0-3 |  | 46
  Grade 3 Loss of appetite, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Grade 3 Loss of appetite, Dose 2, Days 0-3 |  | 0
  Related Loss of appetite, Dose 2, Days 0-3: number analyzed (Participants) | 0 | 166
  Related Loss of appetite, Dose 2, Days 0-3 |  | 32
  Any Drowsiness, Dose 1, Days 0-7 | 52 | 70
  Grade 3 Drowsiness, Dose 1, Days 0-7 | 2 | 0
  Related Drowsiness, Dose 1, Days 0-7 | 37 | 53
  Any Fever, Dose 1, Days 0-7 | 17 | 6
  Grade 3 Fever, Dose 1, Days 0-7 | 0 | 0
  Related Fever, Dose 1, Days 0-7 | 7 | 1
  Any Irritability, Dose 1, Days 0-7 | 69 | 103
  Grade 3 Irritability, Dose 1, Days 0-7 | 4 | 5
  Related Irritability, Dose 1, Days 0-7 | 48 | 87
  Any Loss of appetite, Dose 1, Days 0-7 | 42 | 48
  Grade 3 Loss of appetite, Dose 1, Days 0-7 | 2 | 2
  Related Loss of appetite, Dose 1, Days 0-7 | 22 | 33
  Any Drowsiness, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Any Drowsiness, Dose 2, Days 0-7 |  | 52
  Grade 3 Drowsiness, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Grade 3 Drowsiness, Dose 2, Days 0-7 |  | 0
  Related Drowsiness, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Related Drowsiness, Dose 2, Days 0-7 |  | 39
  Any Fever, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Any Fever, Dose 2, Days 0-7 |  | 16
  Grade 3 Fever, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Grade 3 Fever, Dose 2, Days 0-7 |  | 0
  Related Fever, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Related Fever, Dose 2, Days 0-7 |  | 5
  Any Irritability, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Any Irritability, Dose 2, Days 0-7 |  | 84
  Grade 3 Irritability, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Grade 3 Irritability, Dose 2, Days 0-7 |  | 5
  Related Irritability, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Related Irritability, Dose 2, Days 0-7 |  | 62
  Any Loss of appetite, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Any Loss of appetite, Dose 2, Days 0-7 |  | 51
  Grade 3 Loss of appetite, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Grade 3 Loss of appetite, Dose 2, Days 0-7 |  | 1
  Related Loss of appetite, Dose 2, Days 0-7: number analyzed (Participants) | 0 | 166
  Related Loss of appetite, Dose 2, Days 0-7 |  | 32

13. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Up to 1 month post-vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 160 | 189
Participants | 87 | 140

14. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to study end (Month 9)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 160 | 189
Participants | 5 | 2

15. Secondary Outcome: Number of Subjects With New Onset Chronic Ilnesses (NOCI)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: Up to study end (Month 9)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 160 | 189
Participants | 19 | 38

16. Secondary Outcome: Number of Subjects Reporting Rash
Description: Rash assessed included hives, idiopathic thrombocytopenic purpura and petechiae.
Time Frame: Up to study end (Month 9)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 160 | 189
Participants | 16 | 61

17. Secondary Outcome: Number of Subjects Reporting Adverse Events Resulting in Emergency Room (ER) Visits
Description: Among AEs prompting emergency room visits were: infections, injuries, skin diseases and respiratory diseases.
Time Frame: Up to study end (Month 9)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
Number analyzed (Participants) | 160 | 189
Participants | 17 | 32

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 8-day (Days 0-7) post-vaccination period, Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period, SAEs: during the entire study period (from Month 0 up to Month 9).
Arm/Group | GSK 134612 1 Dose Group | GSK 134612 2 Doses Group
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/189
Serious Adverse Events (participants affected / at risk) | 5/160 | 2/189
Other Adverse Events (participants affected / at risk) | 124/160 | 172/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK 134612 1 Dose Group (N=160) | GSK 134612 2 Doses Group (N=189)
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Otitis media (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK 134612 1 Dose Group (N=160) | GSK 134612 2 Doses Group (N=189)
Bronchiolitis (Infections and infestations) | 1 (1) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 42 (42) | 83 (99)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 21 (22)
Erythema (Skin and subcutaneous tissue disorders) | 28 (28) | 62 (88)
Irritability (Psychiatric disorders) | 69 (69) | 127 (191)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (12)
Otitis media (Infections and infestations) | 18 (19) | 37 (39)
Pain (General disorders) | 35 (35) | 69 (96)
Pyrexia (General disorders) | 27 (27) | 59 (70)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 13 (13)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Somnolence (Nervous system disorders) | 52 (52) | 93 (122)
Swelling (General disorders) | 13 (13) | 38 (46)
Teething (Gastrointestinal disorders) | 10 (11) | 18 (18)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 37 (43)
Viral infection (Infections and infestations) | 3 (3) | 11 (11)
Vomiting (Gastrointestinal disorders) | 6 (6) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.